CLINICAL TRIAL: NCT05647642
Title: The Effect of Premedication Methods to be Applied to Prevent Preoperative Anxiety in Patients Who Will be Operated for Breast Cancer, on Postoperative Anxiety and Pain
Brief Title: The Effect of Premedication on Postoperative Pain and Anxiety in Breast Cancer Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda ARI, Doctor, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2022-09/2057
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Female Patients Under the Age of 65 Who Will Undergo Breast Cancer Surgery
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- low dose midazolam: 0,025 mg/kg Midazolam
  Interventions: Drug: Precedex and dormicum
- high dose midazolam: 0,05 mg/kg Midazolam
  Interventions: Drug: Precedex and dormicum
- low dose dexmedetothymidine: 0.5 mg/kg dexmedetothymidine 10 minute infusion
  Interventions: Drug: Precedex and dormicum
- high dose dexmedetothymidine: 1mg/kg dexmedetothymidine 10 minute infusion
  Interventions: Drug: Precedex and dormicum

INTERVENTIONS:
Drug: Precedex and dormicum — Premedication

SUMMARY:
In this study, it was investigated whether the premedication drug administered before the surgery had an effect on postoperative pain and anxiety scores in female patients under the age of 65 who will undergo breast cancer surgery.

DETAILED DESCRIPTION:
In this study, it was investigated whether the premedication drug administered before the surgery had an effect on postoperative pain and anxiety scores in female patients under the age of 65 who will undergo breast cancer surgery. The STAI-1(State Trait Anxiety İnventory ) form and APAIS (Amsterdam Preoperative Anxiety and İnformation Scale) scale were filled in for all preoperative patients. Afterwards, the patients were treated with either midazolam or dexmedetothymidine, depending on the anesthesiologist's preference. After administration, he was taken to surgery. As intraoperative analgesics, 2 mg/kg tramadol and 15 mg/kg paracetamol were administered to all patients. postoperative recovery time (aldrete 10), 1., 2.,6.,12.,24. VAS score, postoperative nausea-vomiting scale, STAI-1(State Trait Anxiety İnventory ) form, first need time if postoperative analgesic was needed, and 24-hour total analgesic consumption were recorded. It was aimed to examine the effects of different premedications on postoperative pain and anxiety

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2-3
* 18-65 aged
* Female patients

Exclusion Criteria:

* Under 18 years old and over 65 years old
* Having a history of cerebrovascular disease illiteracy
* Have visual and auditory problems İnability to cooperate with cognitive function test
* Having emergency surgery
* Those who are unable to read, understand and sign the consent form
* Patients deemed unsuitable by the investigator

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA 1-2-3, female patients aged 18-65 who will undergo breast cancer surgery
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10-16 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
effect of premedication on postoperative pain and anxiety scores | November 2022-December 2022

CONTACTS AND LOCATIONS:
Locations (1):
- AbdurrahmanYAOTRH, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided